CLINICAL TRIAL: NCT02678481
Title: MR-targeted vs. Random TRUS-guided Prostate Biopsy in Patients With High PSA Values and Previous Negative Biopsy Results: A Randomized Controlled Trial
Brief Title: MR-targeted vs. Random TRUS-guided Prostate Biopsy
Acronym: Pro-Cure2014
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro-Cure PCa 2014
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Prostate Cancer
Keywords: multiparametric magnetic resonance imaging; MR-targeted prostate biopsy; saturation TRUS-guided prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MR-targeted biopsy (Experimental): Patients of arm A receive a targeted MR-guided in-bore prostate biopsy. From each prostate lesion defined in the diagnostic multiparametric MR imaging two targeted biopsy cores will be taken.
  Interventions: Device: MR-guided in-bore prostate biopsy
- TRUS-guided biopsy (Experimental): Patients of arm B receive a saturation TRUS-guided prostate biopsy.
  Interventions: Device: TRUS-guided prostate biopsy

INTERVENTIONS:
Device: MR-guided in-bore prostate biopsy — 2 targeted biopsy cores from each prostate lesion detected at multiparametric MR imaging
  Arms: MR-targeted biopsy
Device: TRUS-guided prostate biopsy — 24-28 systematic biopsy core (saturation scheme)
  Arms: TRUS-guided biopsy

SUMMARY:
To compare prostate cancer (PCa) detection rate of magnetic resonance (MR)-targeted biopsy and transrectal ultrasound (TRUS)-guided biopsy in patients with high PSA values and at least one previous negative prostate biopsy. Subjects will be submitted to a multiparametric MR scan of the prostate and subsequently patients with a suspicious MR for PCa presence will be randomized (1:1) into the two study arms.

DETAILED DESCRIPTION:
In men with previously negative prostate biopsy and persistent elevated PSA value, it is unclear which biopsy strategy offers the highest detection rate for significant PCa. The hypothesis of this study is that MR-targeted biopsy improves the detection rates of significant prostate cancers compared with systematic TRUS-guided prostate biopsy.

Men with at least one previously negative TRUS-guided biopsy and persistently elevated PSA values (> 4 ng/ml) will be submitted to a multiparametric MR imaging examination of the prostate. Subsequently, participants with suspected regions at MR imaging will be randomized (1:1) into the two study arms. In study arm A patients will be submitted to MR-targeted in-bore prostate biopsy based on the multiparametric MR imaging findings. In study arm B patients will be submitted to systematic TRUS-guided prostate biopsy with saturation scheme.

ELIGIBILITY:
Inclusion Criteria:

* men aged 50-80
* at least one negative TRUS-guided prostate biopsy
* PSA > 4 ng/ml
* at least one suspected region detected at multiparametric MR imaging
* signed informed consent

Exclusion Criteria:

* known prostate cancer diagnosis
* contraindication against MR imaging or uncooperative patients

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Prostate cancer detection rate | within the 3 months after MR imaging

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Regge, MD, Principal Investigator — Fondazione del Piemonte per l'Oncologia
Locations (1):
- Fondazione del Piemonte per l'Oncologia - Candiolo Cancer Institute, Candiolo, Turin, Italy

IPD SHARING:
Plan to Share IPD: No